CLINICAL TRIAL: NCT02428621
Title: Prospective Multicentric, Open-label, Randomized Study Assessing the Efficacy of the Removable and Adjustable Preformed Twicare® Appliance Versus Removable Herbst Appliance Treatment in Class II Malocclusion
Brief Title: Early Treatment for Class II Division 1 Malocclusion With Twicare® and Herbst Removable Appliances
Acronym: EffTwicare
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the study is discarded by the sponsor.
Sponsor: FCI System (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-A01629-38
Record Dates: First submitted 2015-04-21; First posted 2015-04-29 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Malocclusion, Angle Class II, Division 1
Keywords: early orthodontic treatment; activator; removable appliance; Twicare®; Herbst appliance
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Twicare® appliance (Experimental): Group treated with the Twicare® appliance. This appliance is a removable mandibular propulsive adjustable preformed medical device. It is made out of soft and stiff thermoplastics. Its two gutters are linked to each other according to different antero-posterior positions. It is EC marked since 2011.
  Interventions: Device: Twicare® appliance
- Removable Herbst appliance (Active Comparator): Group treated with the removable Herbst appliance. This appliance is a medical device measured made composed of telescopic metallic hinges and resin gutters made-to-measure based on dental impression.
  Interventions: Device: Removable Herbst appliance
- Untreated (No Intervention): Children will not wear any interceptive activator. They will have a routine follow-up with their orthodontist waiting for the placing of a fixed appliance.

INTERVENTIONS:
Device: Twicare® appliance — Early orthodontic treatment with the Twicare®. The Class II treatment is initiated at the age of 7-12 years and continued as long as the Class I is achieved.
  The Twicare® is adjusted in mandibular protraction based on the 2/3 of the condylar test and was were worn during 12 to 14 hours a day (at least 4 hours during the day and all night).
  Arms: Twicare® appliance
Device: Removable Herbst appliance — Early orthodontic treatment with the removable Herbst appliance. The Class II treatment is initiated at the age of 7-12 years and continued as long as the Class I is achieved.
  The Herbst appliance is adjusted in mandibular protraction based on the 2/3 of the condylar test and was were worn during 12 to 14 hours a day (at least 4 hours during the day and all night).
  Arms: Removable Herbst appliance

SUMMARY:
The aim of this prospective, multicentric, randomized, open-label study is to assess the efficacy of the removable Twicare® as mandibular propulsive appliance in children aged from 7 to 12 years old in the course of their orthodontic treatment, showing its noninferiority with the removable Herbst. One untreated group will be included to control the internal validity of the study as recommend in noninferiority trials. Patients will have a follow-up every two months during 6 to 12 months as planned in routine care.

DETAILED DESCRIPTION:
A large number of functional appliances, mandibular advancement activators with various designs, fixed or removable, are used in Class II malocclusion correction; one of the largest means being used is the Herbst. These appliances can be individualized, made to measure by the prosthetist or standardised (on market). A new medical device, EC marked and marketed since 2011, the Twicare®, can be used as positioner, growth activator, but also for lingual re-education.

There are numerous publications comparing the activators' effects or the appliance effects on mandibular growth, but none have studied the Twicare®. The aim of this study is to assess the efficacy of this specific removable appliance in mandibular advancement in Class II skeletal in children aged from 7 to 12 years old. The appliance will be compared with the Herbst and one untreated group will be included to control the internal validity of the study as recommend in noninferiority trials.

Patients will have a follow-up every two months during 6 to 12 months until the Class I occlusion is achieved. A lateral cephalogram and a dental silicon impression will be performed at the beginning (T0) and at the end of the treatment (T1) in order to evaluate cephalometric measurement changes, ANB, overjet and canine and molar class evolutions. The data collected at the beginning and at the end of the treatment will be analyzed and compared aware from patient, treatment and time, in order to assess the Twicare® noninferiority compared to the Herbst and to confirm the superiority of these two appliances versus observation. We will study, in parallel, the nasal ventilator function as well as comfort, compliance, tolerance and acceptability of the device via an auto-questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Children with Class II division 1 malocclusion
* Overjet ≥ 4 mm,
* ANB > 4°,
* Good cooperation (motivation and good dental hygiene),
* Incisors width compatible with the available Twicare® appliance sizes, according to the manufacturer recommendations.
* Written Informed Consent of the Child,
* Affiliated to health insurance,
* Parents able to receive informed consent and to express their approval for their child to take part in this investigation.

Exclusion Criteria:

* Non well-balanced periodontal disease,
* Temporal-mandibular dysfunction,
* Severe bruxism noctural episodes,
* Known allergy or intolerance to one of the activators' components.
* Foreseeable follow-up difficulties,
* Minor under guardianship,
* Simultaneous participation to an interventional study.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2015-07; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
A point-nasion-B point (ANB) angle change | 6-12 months
  ANB change is measured in lateral cephalograms between the beginning (T0) and the end (T1) of the treatment.

SECONDARY OUTCOMES:
Overjet change using dental silicone impression | 6-12 months
  Assessment of the overjet change between the beginning (T0) and end (T1) of the treatment using dental silicone impression.
Cephalometric analysis (Tweed analysis of lateral cephalograms) | 6-12 months
  Assessment of cephalometric measurement changes between T0 and T1 based on Tweed analysis of lateral cephalograms: the lower and upper incisor inclination (I/APog and i/APog) and mandibular corpus growth increase will be investigated in particular.
Nasal ventilation (Peak Nasal Inspiratory Flow (PNIF) change) | 6-12 months
  Assessment of the Peak Nasal Inspiratory Flow (PNIF) change between T0 and T1. The PNIF is measured with a spirometer.
Treatment acceptability (subjective) | 6-12 months
  Subjective assessment of the appliance wearing compliance and treatment tolerance/acceptability with auto-questionnaire and filling up of a diary (wearing timesheet).
Compliance (appliance wearing based on patient interview with a questionnaire.) | 6-12 months
  Clinical Assessment of appliance wearing based on patient interview with a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Renaudin, Dr, Principal Investigator — Department of Othodontics, Faculty of Dentistry, University of Nantes, Nantes, France
Locations (3):
- France (3):
  - Orthodontic Private Center, Cherbourg
  - Department of Orthodontics, Faculty of Dentistry, Nantes
  - Department of Orthodontics, Faculty of Dentistry, Rennes

REFERENCES:
- See also: Twicare® appliance — http://www.medventiv.com/index_en.php